CLINICAL TRIAL: NCT05852639
Title: Fetal Cerebroplacental Ratio at Term for Prediction of Adverse Neonatal Outcome in Pregnancies Complicated by Gestational Diabetes
Brief Title: Fetal CPR at Term for Prediction of Adverse Neonatal Outcome in Pregnancies Complicated by GDM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mariam Alaaeldin Aly Gabr, Dr., Cairo University
Other Study IDs: MD-329-2022
Record Dates: First submitted 2023-05-02; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Gestational Diabetes
Keywords: cerebroplacental ratio; adverse neonatal outcome
MeSH Terms: conditions — Diabetes, Gestational | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Insulin: patients on insulin treatment for gestational diabetes
  Interventions: Device: Ultrasound
- Metformin: patients on metformin treatment for gestational diabetes
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Routine obstetric ultrasound will be done at term (at 37 weeks gestation): to confirm gestational age, assess fetal weight and amniotic fluid index and to exclude fetal anomalies.Doppler study and cerebroplacental ratio assessment will be done at 37 weeks gestation and repeated every two weeks

SUMMARY:
The goal of this observational study is to evaluate fetal cerebroplacental ratio at term and its relation to adverse neonatal outcome in patients with gestational diabetes. The main question[s] it aims to answer are:

* To evaluate the efficacy (sensitivity & specificity) of fetal cerebroplacental ratio at term in prediction of adverse neonatal outcome in pregnancies complicated by gestational diabetes
* To evaluate the difference in fetal cerebroplacental ratio in patients treated by insulin & those on metformin
* to evaluate the incidence of adverse neonatal outcome in patients treated by insulin & those on metformin.

Participants will undergo ultrasound and doppler study at 37 weeks & every two weeks thereafter till delivery. Neonatal assessment will be done after delivery to exclude adverse outcomes.

DETAILED DESCRIPTION:
pregnant females in the reproductive age, pregnant ≥37 weeks, who were diagnosed with gestational diabetes by routine screening at 24-28 weeks, and are on metformin or insulin treatment. Informed consent, to share in the study, will be taken from all participants after describing the aim of the study and the potential hazards.

The patients enrolled in our study will be divided into two equal groups according to their treatment regimens:

(Group A): 130 patients who are on insulin treatment

(Group B): 130 patients who are on metformin

*All participants will be subjected to the following:

A) Full history taking:

Including personal, menstrual, obstetric, present, past & family history. B) Complete Physical Examination (general & local).

C) Investigations:

* Routine baseline investigations:

  1. Complete blood picture, Rh typing, liver & kidney functions.
  2. HbA1C estimation.
  3. Surveillance of maternal diabetes: daily fasting and 2- hour postprandial capillary glucose measurement.
  4. Routine obstetric ultrasound will be done at term (at 37 weeks gestation): to confirm gestational age, assess fetal weight (EFW) and amniotic fluid index (AFI) and to exclude fetal anomalies.
* Doppler ultrasonography assessment:

Doppler study and Cerebroplacental ratio assessment will be done at 37 weeks gestation and repeated every two weeks.To reduce inter-operator variability, a single experienced sonographer will perform all sonograms.

The mode of delivery and the gestational age at delivery will be noted

Early neonatal assessment:

1. 1&5 minutes APGAR score
2. Neonatal blood glucose
3. Neonatal cord blood PH
4. The need for NICU admission

ELIGIBILITY:
Inclusion Criteria:

* Maternal age: 18-40 years
* Diagnosed with gestational DM and are on insulin or metformin treatment.
* Single living pregnancy.
* Gestational age ≥ 37 weeks (confirmed by a reliable date for the last menstrual period and 1st trimester ultrasound scan).

Exclusion Criteria:

* Fetal anomalies.
* Maternal chronic diseases esp. renal disease, epilepsy or CNS lesion.
* Pregnancy induced medical disorders.
* IUGR (EFW below the 10th percentile for gestational age).
* Rupture of membranes or oligohydramnios (AFI < the fifth percentile).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients in our study will be recruited from Kasr al-Ainy hospital inpatient departments as follows: pregnant females in the reproductive age, pregnant ≥37 weeks, who were diagnosed with gestational diabetes by routine screening at 24-28 weeks, and are on metformin or insulin treatment.
Sampling Method: Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2022-11-30 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy (sensitivity & specificity) of fetal cerebroplacental ratio at term in prediction of adverse neonatal outcome in pregnancies complicated by gestational diabetes | 17 months

SECONDARY OUTCOMES:
To evaluate the difference in fetal cerebroplacental ratio in both groups | 17 months
To evaluate the incidence of adverse neonatal outcome in both groups | 17 months

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Gabr, Principal Investigator — Cairo University
Locations (1):
- Kasr al-ainy hospital, Faculty of Medicine - Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided